CLINICAL TRIAL: NCT06959212
Title: Investigation of Mnesic Capacities in Patients With a Disorder of Consciousness - MemoDoC
Brief Title: Investigation of Mnesic Capacities in Patients With a Disorder of Consciousness
Acronym: MemoDoC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut du Cerveau et de la Moelle (ICM Institute) (Unknown); Sorbonne University, Paris, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP240232
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Disorders of Consciousness
Keywords: DoC; hidden cognition; subjective experience; memory; neurophysiology
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients suffering or who have suffered from a Disorder of Consciousness (Experimental)
  Interventions: Other: Physiological recordings, Semi-structured interviews, Psychological scales
- Conscious Patients treated in Intensive Care Unit (Active Comparator)
  Interventions: Other: Physiological recordings, Semi-structured interviews, Psychological scales

INTERVENTIONS:
Other: Physiological recordings, Semi-structured interviews, Psychological scales — (Neuro)-physiological paradigms based on EEG, ECG, electrodermal activity, and respiratory activity recordings, and auditory and olfactive stimuli, to assess memory processes without the need to communicate ('no report' approach) in patients suffering from a Disorder of Consciousness and conscious controls. Semi-structured interviews and neuropsychological assessments (scales) in patients who have recovered from a Disorder of Consciousness and conscious controls to explore memories and subjective experience of the ICU

SUMMARY:
Following severe brain damage, some individuals lose partial or total awareness of themselves and their environment, falling into a coma that can evolve towards a Disorder of Consciousness (DoC). Accurately diagnosing the depth of consciousness alteration, and thus characterizing the patient's residual state of consciousness, is a real medical challenge, yet crucial for establishing a neurological prognosis, predicting cognitive outcome, and guiding medical decisions. Clinicians attempt to classify DoC patients into different global states (e.g. coma, Unresponsive Wakefulness Syndrome (UWS), Minimally Conscious State (MCS)) depending on their residual level of arousal and awareness.

In recent years, the improvement of diagnostic tools and the use of a multimodal approach combining clinical, neurophysiological and neuroimaging examinations, have greatly refined this assessment and revealed the existence of possible discrepancies between clinical observation (e.g. poor consciousness state like UWS) and brain activity (richer, MCS+ type, or even conscious) so-called Cognitive-Motor Dissociation, making it essential to search for any 'hidden cognition' not revealed by the clinical behavioral examination. It is therefore essential to have tools that can not only probe consciousness level, but also provide a detailed profile of patients' residual cognitive abilities - such as language, attention or memory - which are essential dimmensions of conscious experience and shape waking cognitive life. This could crucially improve the neurological diagnostic and prognostic' accuracy of these disorders, as well as allowing to infer the eventual subjective experience of these patients. Indeed, we still know very little about the possible conscious 'contents' involved in these states. What does the possible 'mental life' of DoC patients look like? A multidimensional exploration of their cognition is needed, requiring the development of innovative methods capable of probing cognitive functions in the absence of any communication with the patient.

Thus, the general aim of this study lies in the development of tools for the cognitive exploration of DoC patients and their application at patients' bedside in the Intensive Care Unit (ICU). We're particularly interested in assessing memory capacities in these patients, as exploration of memory has immediate clinical implications, since memory encoding during DoC could impact patients' quality of life and be implicated in the occurrence of post-traumatic stress disorder (PTSD) in case of consciousness recovery. More specifically, we want to tackle the following questions: Are patients suffering from a DoC able to form, consolidate and retrieve new memories (anterograde memory)? Are they able to recall memories from their 'past life' (retrograde memory)? Previous research suggests that some DoC patients retain the ability to reactivate old autobiographical memory traces, and to present automatic short-term sensory memory processes, or residual working memory. Nevertheless, DoC patients' memory abilities have been little studied to date, despite their clinical relevance.

We postulate that memory could be differentially preserved between different clinical states of DoC such as UWS and MCS. At the group level, we expect MCS patients to have better learning and memory retrieval abilities than UWS patients. We therefore expect memory functions to be affected by brain lesions and, consequently, by consciousness alteration, although we envisage the preservation of unconscious memory processes (e.g. in non-declarative memory subtypes such as perceptual memory) in UWS patients. We hypothesize that the presence of robust markers of memory processes will vary, at the single-patient level, according to the types and stages of memory tested, informing the cognitive profile of the patient suffering from a DoC.

By providing information on the potential presence of memory capacities that cannot be revealed by clinical examination, the physiological tools we are developing in this study will open a crucial window onto non-communicating patients' cognition. Defining DoC patients' memory profile could not only improve their care during and after the disorder (reflection on the quality of life in ICU; better understanding of cognitive and psychological symptoms occurring after a DoC (e.g. amnesia, PTSD); orientation of rehabilitation strategies), but also improve the diagnostic accuracy of these troubles if memory proves to be differentially preserved between different DoC states such as UWS and MCS. Ultimately, we aim to refine the neurological prognosis of these non-responsive patients, by predicting their cognitive outcome thanks to these innovative physiological tools. On a more fundamental level, this project questions the interplay of memory and consciousness, exploring which forms of memory do and do not require a conscious state.

DETAILED DESCRIPTION:
This study investigates the memory capacities of Intensive Care Unit patients suffering from a Disorder of Consciousness (DoC) resulting from severe brain injury. Given the complexity of human memory, this study was designed to provide a nuanced profile of mnesic abilities by examining various types, stages, and temporal dimensions of memory. Specifically, the protocol targets progressively complex types of memory-perceptual, episodic, and autobiographical-alongside two key stages: encoding and retrieval. It also considers two temporal perspectives: (1) memory processes during the DoC (assessed indirectly through physiological markers) and (2) memory retrieval after the DoC, in patients who regain consciousness (assessed directly through subjective reports).

1. We first aim to identify robust and specific physiological markers of memory processes occurring during the period of altered consciousness in the ICU. To this end, we developed two auditory protocols using high-density electroencephalography (hdEEG) and electrocardiography (ECG) to assess the formation of new memories in non-communicating DoC patients (1a; anterograde memory). These protocols focus on two types of memory: perceptual memory, which enables the storage and interpretation of sensory information (e.g., recognition of the sounds of the artificial respirator or the voices of caregivers), and episodic memory, which allows individuals to recall specific events within their context (e.g., family visits, painful procedures) and serves as a foundation for autobiographical memory which supports the sense of identity. In practice, these protocols are conducted over two consecutive days in the ICU: Day 1 is dedicated to the putative encoding of new memories through exposure to specific auditory stimuli, while Day 2 assesses their long-term retrieval using 'old-new' paradigms, which contrast brain responses to stimuli presented on Day 1 ('old') with responses to novel stimuli introduced only on Day 2 ('new'). We also developed a complementary protocol based on hdEEG, ECG and electrodermal and respiratory activity recordings, using auditory and olfactory stimuli, to investigate the retrieval of past autobiographical memories (1b; retrograde memory), that is memories from the patient's life prior to the onset of the disorder.
2. In parallel with this detection of implicit physiological correlates of memory, we will also employ a direct approach in patients who have emerged from a DoC. Using semi-structured interviews, we will gather explicit evidence of their subjective experiences and memories of the period of impaired consciousness. These may include internal conscious experiences (e.g., memories of dreams, hallucinations, emotions, or thoughts), external conscious experiences (e.g., family visits, painful procedures), as well as memories related to stimuli from experimental paradigms (e.g., auditory cues presented during physiological recordings) and memories of a musical memory probe played during the DoC. These interviews will be accompanied by neuropsychological tests assessing overall memory and cognitive functioning and the occurrence of PTSD.

We will apply supervised machine learning techniques, including classification methods, to detect the presence or absence of memory processes at the individual patient level, based on predefined mnesic markers used as evaluation criteria. In parallel, we will conduct second-order analyses, involving group-level comparisons between DoC patients and conscious ICU control patients, as well as between subgroups of DoC patients (e.g., UWS vs. MCS patients; focal vs. diffuse etiologies). These comparisons will be carried out using permutation statistics, statistical modeling, and/or parametric or non-parametric tests (e.g., Student's t-test, Wilcoxon-Mann-Whitney test).

ELIGIBILITY:
Inclusion criteria

Patients suffering from a Disorder of Consciousness:

* Patient not conscious according to the CRS-R scale (Kalmar & Giacino, 2005)
* Age over 15 years and 3 months
* Free and informed consent signed by a third party (parental authority, trusted support person)

Conscious patients (controls) :

* Age over 15 years and 3 months
* Cared for in an Intensive Care Unit
* Free and informed consent signature

Patients who have regained consciousness after having suffered from a Disorder of Consciousness (if not included during their disorder):

* Age over 15 years and 3 months
* Free and informed consent signature if able, otherwise signature of relative (holders of parental authority for minors)
* Patient who has been unconscious for at least 3 days according to the CRS-R scale Exclusion criteria: - Deep sedation (Intracranial hypertension, refractory status epilepticus)
* Previous severe neurodegenerative disease (e.g. Alzheimer's disease, Lewy body dementia)
* Deafness
* Patients under guardianship or trusteeship
* Pregnant and breast-feeding women

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
EEG-Electrodermal activity | during hospitalization and at a distance during a post-resuscitation follow-up consultation for the second semi-structured interview assessing the recovery of the musical memory probe, generally between 3 and 12 months
  Composite primary outcome measure: Presence of at least one of the following three predifined markers of memory processes:
  * EEG cognitive evoked potentials
  * Significant modulation of electrodermal activity
  * Evidence of recollection of an auditory memory probe delivered during the Disorder of Consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Rohaut, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - APHP, Pitié-Salpêtrière Hospital, Department of Anesthesia and Intensive Care, NeuroSurgery ICU, Paris
  - APHP, Pitié-Salpêtrière Hospital, Department of Neurology, Neuro-ICU, Paris

IPD SHARING:
Plan to Share IPD: No